CLINICAL TRIAL: NCT01443338
Title: A Phase4,Multicenter, Randomized,Double-blind,Double Dummy, Parallel Controlled Study Evaluating the Efficacy and Safety of Triptergium Wilfordii and Acitretin in Treatment of Chinese Patients With Moderate to Severe Psoriasis Vulgaris
Brief Title: Study Evaluating the Efficacy and Safety of Triptergium Wilfordii and Acitretin in Psoriasis Vulgaris - CHINA201002016-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Min Zheng, Head of dermatology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHINA201002016-2
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Triptergium wilfordii; Acitretin; psoriasis vulgaris
MeSH Terms: interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptergium Wilfordii (Active Comparator): a kind of traditional chinese medicine
  Interventions: Drug: Triptergium Wilfordii
- Acitretin (Active Comparator)
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Triptergium Wilfordii — Tablet,10mg/Tab,20mg Tid,No more than 8 Weeks
  Arms: Triptergium Wilfordii
Drug: Acitretin — Capsule,10mg/Cap,30mg Qd,no more than 8 weeks
  Arms: Acitretin

SUMMARY:
The purpose of this study is to determine whether Triptergium wilfordii, and Acitretin are effective and safe in the treatment of patient of moderate to severe psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, between the age 18 and 75 years.
* Have a diagnosis of psoriasis vulgaris,PASI score of 7 or greater.
* Capable of giving informed consent and the consent must be obtained prior to any study related procedures.

Exclusion Criteria:

* Currently have erythrodermic,guttate or pustular psoriasis.
* Have any active dermatoses which may affect disease assessment of psoriasis.
* Have used any investigational drug,any biologic or any systemic immunosuppressants within the previous 1 month..
* Have used topical medications/treatments that could affect psoriasis or PASI evaluation (eg, corticosteroids, tar, phototherapy et al.) within 2 weeks.
* Have any acute or chronic or recurrent infectious disease,which was difficult to control.
* Have the history of HBV or HCV infection,or HIV antibody test positive.
* AST, ALT or blood fat levels must be within 1.5 times the ULN range for the laboratory conducting the test.
* Are pregnant, nursing, or planning pregnancy in the coming two years(both men and women) while enrolled in the study.
* Have any severe systemic disease or have a history of malignancy.
* Have shown a previous hypersensitivity to Triptergium wilfordii or Acitretin.
* Have any other condition not suitable to join in trial,which are judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plaque psoriasis as assessed by PASI(psoriasis area and severity index) response or PASI 75 (a patient that has an improvement from baseline PASI of at least 75%) | to 8 weeks treatment

SECONDARY OUTCOMES:
Change from baseline in plaque psoriasis as assessed by PASI response or PASI 50 (a patient that has an improvement from baseline PASI of at least 50%) | to 8 weeks treatment
Change from baseline in plaque psoriasis as assessed by PASI response or PASI 90 (a patient that has an improvement from baseline PASI of at least 90%) | to 8 weeks treatment
Laboratory parameters, rates of AEs, and percentage of patients requiring interruption or discontinuation of study drug due to AEs | to 8 weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China